CLINICAL TRIAL: NCT04899856
Title: Randomized Study of TransAeris® System for Enhanced Recovery After Surgery (ERAS) in Cardiac Surgery Patients at Risk of Prolonged Mechanical Ventilation
Brief Title: Randomized Study of TransAeris® System in Cardiac Surgery Patients at Risk of Prolonged Mechanical Ventilation
Acronym: ERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-1000-105
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Ventilator Induced Diaphragm Dysfunction
Keywords: VIDD

STUDY DESIGN:
Intervention Model Description: This study is an open label, randomized, cross-over study in adult open cardiac surgery patients. All subjects will receive TransLoc electrodes at the time of open sternotomy cardiac procedure. Half of subjects will have TransAeris turned on upon entry to ICU, the other half will receive standard of care with TransAeris turned on if still intubated on mechanical ventilation after 120 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control / Crossover to TransAeris Therapy (Other): The "Control" group will be treated per standard hospital policy following electrode implant. If the participant is not liberated from mechanical ventilation after 120 hours (5 days), the participant will begin using TransAeris therapy. The participant will use the study device in the ICU until liberated from the ventilator but no longer than 30 days after implant surgery.
  Interventions: Device: TransAeris
- Treatment with TransAeris Therapy (Experimental): The "Treatment" group will start TranAeris therapy shortly after arrival in the Intensive Care Unit (ICU). Participants will use the study device in the ICU until liberated from the ventilator but no longer than 30 days after implant surgery.
  Interventions: Device: TransAeris

INTERVENTIONS:
Device: TransAeris — TransAeris is used to provide neuromuscular electrical stimulation to the diaphragm while the patient is on mechanical ventilation to prevent, slow, or reverse diaphragm disuse atrophy and, more generally, to prevent and treat VIDD.

SUMMARY:
This study will be conducted as a randomized trial of the TransAeris system for the prevention and treatment of ventilator-induced diaphragm dysfunction (VIDD) in patients identified prior to surgery to be at greater risk of prolonged mechanical ventilation (PMV).

DETAILED DESCRIPTION:
This study is an open label, randomized, cross-over study in adult open cardiac surgery patients. All subjects will receive TransLoc electrodes at the time of open sternotomy cardiac procedure. Half of subjects will have TransAeris turned on upon entry to ICU, the other half will receive standard of care with TransAeris turned on if still intubated on mechanical ventilation after 120 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing an open cardiac procedure by median sternotomy
2. Subject is at risk of prolonged mechanical ventilation according to one or more of the following criteria:

   * Prior open cardiac surgery
   * Left Ventricular Ejection Fraction (LVEF) ≤ 30%
   * History of TIA or CVA
   * Pre-operative or anticipated intraoperative intra-aortic balloon pump
   * History of COPD
3. Subject is at least 22 years of age
4. Informed consent has been obtained from the patient

Exclusion Criteria:

1. Subject is on invasive mechanical ventilation prior to procedure
2. Subject has known or pre-existing phrenic nerve paralysis
3. Subject is having a left ventricular assist device implanted
4. Subject has progressive, non-reversible neuromuscular disease affecting the diaphragm
5. Subject is pregnant or lactating
6. Subject is actively participating in another clinical study which could affect outcomes in this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experiencing serious device-related adverse effects | 60 days after implantation
  All participants will be assessed for serious device-related adverse effects
Proportion of subjects weaned at 48 hours and 120 hours | 90 days after study completion
  Time on mechanical ventilation will be compared between the Control and Treatment groups

SECONDARY OUTCOMES:
Number of subjects experiencing device-related adverse events | 90 days after study completion
  All participants will be assessed for device-related adverse events
Average number of days in the Intensive Care Unit (ICU) | 90 days after study completion
  Time in the ICU will be tracked for all study participants and averaged
Average number of days in the hospital | 90 days after study completion
  Time in the hospital will be tracked for all study participants and averaged

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P Onders, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] David CH, Vourc'h M, Guimbretiere G, Mugniot A, Lacoste P, Cadiet J, Rozec B, Arora R, Pelletier M, Sabik J, Onders R. Multicentre Study of Diaphragm Pacing in High-Risk Cardiac Surgery to Decrease Postoperative Mechanical Ventilation. Eur J Cardiothorac Surg. 2026 Jan 6;68(1):ezaf472. doi: 10.1093/ejcts/ezaf472. PMID 41416899